CLINICAL TRIAL: NCT02091102
Title: Evaluation of the Safety and Efficacy of the Pico Laser With a Specialized Lens Array for the Treatment of Wrinkles
Brief Title: Evaluating the Safety and Efficacy of the Pico Laser With a Specialized Lens Array for the Treatment of Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN13-PICO-LENS-DM
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Wrinkles
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 755nm Alexandrite Laser (Experimental): 755nm Alexandrite Laser
  Interventions: Device: 755nm Alexandrite Laser

INTERVENTIONS:
Device: 755nm Alexandrite Laser — 755nm Alexandrite Laser for the treatment of Wrinkles

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the treatment of wrinkles using a 755nm Alexandrite Laser.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy non-smoking (must have quit 6 months prior) male or female between 18 and 65 years old.
2. Is willing to consent to participate in the study.
3. Is willing to comply with all requirements of the study including biopsies, being photographed, following post treatment care and attending all treatment and follow up visits.

Exclusion Criteria:

1. The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. The subject is hypersensitive to light exposure OR takes photo sensitized medication.
3. The subject has active or localized systemic infections.
4. The subject has a coagulation disorder or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy {greater than 81 mg per day}).
5. The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 3 months prior to entering this study.
7. The subject has used Retin A or Accutane within 6 months prior to enrollment.
8. The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
9. The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
10. The subject has a history of keloids.
11. The subject has evidence of compromised wound healing.
12. The subject has a history of squamous cell carcinoma or melanoma.
13. The subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications or has an autoimmune disorder.
14. The subject has an allergy to lidocaine and epinephrine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McDaniel Institute of Anti Aging Research, Virginia Beach, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 755nm Alexandrite Laser
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 19
  Race/Ethnicity: Hispanic | 1
Fitzpatrick Skin Type Score [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    I | 4
    II | 15
    III | 1
    IV | 0
    V | 0
    VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Photographic Evaluation of Wrinkle Severity at Baseline
Description: Blinded evaluators grade photographs using the Fitzpatrick wrinkle severity scale and provide an overall score for each timepoint. The Fitzpatrick wrinkle scale classifies wrinkles on a scale from 1 (mild) to 9 (severe). Scores of 1-3 are for mild wrinkles, meaning that there are fine texture changes with subtly accentuated skin lines. Scores of 4-6 are for fine to moderate depth wrinkles or moderate amount of lines with distinct popular elastosis and dyschromia. Scores of 7-9 are for fine to deep wrinkles, with numerous lines with or without redundant skin folds. It is characterized by multiple papules and confluent elastosis.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 20
score on a scale | 5.25 (.851)

2. Primary Outcome: Photographic Evaluation of Wrinkle Severity at 1 Month Post Last Treatment
Description: as for outcome 1
Time Frame: 1 Month Follow Up Post Last Treatment
Population: One subject was unable to return to clinic for the 1 month visit due to a family emergency.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 19
score on a scale | 4.74 (.991)

3. Primary Outcome: Photographic Evaluation of Wrinkle Severity at 3 Month Follow Up Post Last Treatment
Description: as for outcome 1
Time Frame: 3 Month Follow Up Post Last Treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 20
score on a scale | 4.25 (1.07)

4. Primary Outcome: Photographic Evaluation of Wrinkle Severity at 4 Month Follow Up Post Last Treatment
Description: as for outcome 1
Time Frame: 4 Month Follow Up Post Last Treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 20
score on a scale | 3.9 (1.07)

5. Primary Outcome: Photographic Evaluation of Wrinkle Severity at 6 Month Follow Up Post Last Treatment
Description: as for outcome 1
Time Frame: 6 Month Follow Up Post Last Treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 20
score on a scale | 4 (1.21)

6. Other Pre Specified Outcome: Satisfaction Questionnaire
Time Frame: up to 6 months post last treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse event data were collected up to 6 months post last treatment.
Arm/Group | 755nm Alexandrite Laser
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 19/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 755nm Alexandrite Laser (N=20)
pain (Nervous system disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 17
Edema (Skin and subcutaneous tissue disorders) | 7
Bruising (Skin and subcutaneous tissue disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 3
Dryness (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.